CLINICAL TRIAL: NCT06539663
Title: The Role of OmniLenz® in the Treatment of Small Corneal Perforations Secondary to Exposure Keratitis in ICU Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Farwaniya Hospital (Other Government)
Responsible Party: Principal Investigator, Nancy Lotfy, MD, Associate Professor of Ophthalmology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-632-4385
Record Dates: First submitted 2024-07-30; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Corneal Perforation; Exposure Keratitis; Infectious Keratitis
MeSH Terms: conditions — Corneal Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of Corneal Perforation (Experimental): All patients were prescribed Fortified Vancomycin (50mg %) and Fortified Fortum (50mg %) antibiotic eye drops for initial exposure keratitis with corneal infiltration. Then treatment was modified according to culture and sensitivity results.
  Subsequent corneal perforation developed for which OmniLenz® was applied in all patients for 1 week.
  Interventions: Combination Product: OmniLenz®

INTERVENTIONS:
Combination Product: OmniLenz® — OmniLenz® applied for 1 week in all patients after development of corneal perforation

SUMMARY:
Case series of 5 ICU patients in Farwaniya Hospital who developed exposure keratitis and a subsequent small corneal perforation between April 2022 and April 2024.

The investigators highlight the non-surgical role of OmniLenz® in the treatment of small corneal perforations secondary to exposure keratitis. The inclusion criteria were corneal perforation less than 1mm in size, positive culture & sensitivity results and showing initial improvement on topical antibiotic eye drops.

DETAILED DESCRIPTION:
The primary outcome measures were healing of the corneal perforation, a negative Seidel test and reformation of the anterior chamber.

Secondary outcome measures were improvement of all three of ciliary injection, state of epithelial defect, and corneal infiltration.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* Patients with small corneal perforations measuring < 1 mm in diameter. Those with larger perforations (>1mm) were excluded.
* Patients with conclusive results of keratitis (confirmed via culture and sensitivity scraping) AND showing improved keratitis following antibiotic treatment. Those with no confirmed keratitis through C&S or with inconclusive scraping results were excluded.
* No age or gender restrictions were applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Size of corneal perforation | one week
  Size of corneal perforation will be measured in mm using slit lamp examination

SECONDARY OUTCOMES:
size of epithelial defect | one week
  Size of epithelial defect will be measured in mm using slit lamp examination

CONTACTS AND LOCATIONS:
Locations (1):
- Farwaniya Hospital, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No